CLINICAL TRIAL: NCT03431363
Title: A Pilot Study to Assess the Role of Cannabis Added to the Supportive Care Regimen During Chemoradiation for Head and Neck Cancer
Brief Title: Medical Cannabis During Chemoradiation for Head and Neck Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-8493
Record Dates: First submitted 2017-12-03; First posted 2018-02-13 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (less than 10 mL in an EDTA tube), urine (less than 15 mL), and oral swab samples will be collected from patients at baseline, once during weeks 1-2, once during week 5-6, and at the time of post-treatment follow-up appointments. Blood tests are routinely performed on a weekly basis for patients receiving systemic therapy and all attempts will be made to coordinate biospecimen collection for study purposes with biospecimen collection for standard clinical care in order to minimize patient inconvenience.
  Each specimen will be analyzed in the Stable Isotope & Metabolomics Core Facility of the Diabetes Research Center under the direction of Dr. Irwin Kurland.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Patient dosing options will be stratified into three groups defined as standard, frail/elderly (age > 65 or ECOG 2), and cannabis-experienced (> weekly use of cannabis in the past year outside of NYC Medical Marijuana program). NYC specified cannabis formulation options are defined by THC:CBD ratio as 1:1, low THC:high CBD, high THC:low CBD, and high THC:high CBD.

SUMMARY:
The primary purpose of the study is to observe the adherence and health seeking behavior of patients with Head and Neck cancer (HNC) certified to obtain medically certified cannabis as part of their supportive care regimen undergoing treatment with definitive or adjuvant concurrent chemoradiation (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed squamous cell carcinoma of the head and neck region planned for definitive or adjuvant treatment with concurrent radiation therapy and systemic therapy
* Patients may receive platinum-based chemotherapy or cetuximab concurrently with radiation therapy
* Age >18 years and ECOG performance status <2 (Karnofsky >60).
* Patients must be willing to use medically certified cannabis as directed after study enrollment
* Patients must be able to read English, Spanish, or French fluently
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior diagnosis of cannabis use disorder as defined in the DSM-V
* Current opioid use disorder on maintenance opioid therapy
* Current active use of smoked cannabis or cannabis derivatives AND unwillingness to cease use of non-medically certified cannabis for the duration of study participation.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cannabis derivatives
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck cancer that meet the eligibility criteria as described above
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Patients' adherence to registering for medically certified cannabis | Through study completion, an average of 12 months
  The primary endpoint of aim 1 is a determination of the number of patients registering for medically certified cannabis as assessed as the number (frequency) as well as proportion of patients registering on New York State Medical Marijuana website
Patients' adherence to procuring medically certified cannabis | Through study completion, an average of 12 months
  The primary endpoint of aim 2 is a determination of the number of patients procuring medically certified cannabis as assessed as the number (frequency) as well as proportion of patients obtaining marijuana from dispensary.

SECONDARY OUTCOMES:
Length of time for patients to obtain medically certified cannabis | Through study completion, an average of 12 months
  The primary endpoint of aim 3 is the length of time it takes patients to obtain medically certified cannabis as assessed by the time elapsed in number of days from study enrollment until medically certified cannabis acquisition and use.

CONTACTS AND LOCATIONS:
Overall Officials: Rafi Kabarriti, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No